CLINICAL TRIAL: NCT03123510
Title: Role of Synbiotics on a Weight Loss Intervention Program: Effect on Microbiome
Brief Title: Effect of a Synbiotic Supplement on a High-protein Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Dakota State University (Other)
Collaborators: Sanford Health (Other)
Responsible Party: Principal Investigator, Eduardo Huarte, Assistant Reseacrh Professor, South Dakota State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1604005
Record Dates: First submitted 2017-03-29; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: probiotics; prebiotics; synbiotics; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: One group will receive a synbiotic supplement and the other placebo capsules.
Who Masked: Participant, Care Provider
Masking Description: Neither the volunteers nor the coaches will be aware
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic supplement (Experimental): Bifidobacterium spp plus bimuno- galacto-oligosaccharides
  Interventions: Dietary Supplement: Bifidobacterium spp plus bimuno- galacto-oligosaccharides
- placebo (Placebo Comparator): sugar pills
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium spp plus bimuno- galacto-oligosaccharides — Volunteers will be asked to take one probiotic capsule and one prebiotic satchel daily.
  Arms: Synbiotic supplement
Dietary Supplement: Placebo — Volunteers will be asked to take one placebo capsule and one placebo satchel daily.
  Arms: placebo

SUMMARY:
The objective of the trial is to study how a synbiotic treatment will affect weight loss and management in individuals enrolled in weight loss diet Profile®. The investigators propose to follow up 2 cohorts of Profile® subjects during 6 months. One group will receive a synbiotic treatment supplement (Bifidobacterium spp plus bimuno- galacto-oligosaccharides (B-GOS)) while the other group will receive placebo capsules. Anthropomorphic and metabolic analysis will be performed by-monthly. Fecal samples will be obtained before and after the dietary intervention and samples will be sequenced trough next generation DNA sequencing to analyze the gut microbiota. Because dietary interventions with high protein and low glycemic index have been shown to be effective in reducing weight, but has also been linked to potential colon harm due to increased fermentation of undigested protein on the colon, the investigators expect supplementation of Profile® with a synbiotic product will lead to an increased overall wellbeing without compromising weight management.

DETAILED DESCRIPTION:
The investigators intend to recruit 40 new Profile® members and to randomly divide them into 2 groups; Group A will follow the conventional coaching and diet plan, while group B will also receive a daily dose of the synbiotic treatment (group A will receive a placebo supplement similar in appearance and caloric content to the synbiotic treatment). Volunteers will be followed for 6 months, and weight loss, waist circumference, BMI and glucose and cholesterol levels will be assessed monthly. Dual-energy x-ray absorptiometry (DXA) will be used to analyze body composition at the beginning and end of the dietary interventions. Fecal samples will be obtained at the beginning and the end of the study. Because both our pre- and probiotic supplements have been reported to increase the concentration of satiating bacteria-derived metabolites, we expect that the individuals on the group B (synbiotic supplement) will experience a higher weight loss as well as more significant drops in glucose and cholesterol levels. Because synbiotic treatments have been reported to facilitate GI passage, the investigators expect volunteers in group B will also report improved bowels movements and general wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Any individual aged 18-80 years participating in the Profile weight loss/management diet

Exclusion Criteria:

* Pregnant
* Requires special diets or dietary regimens
* On long term antibiotic therapy
* Diagnosed with gastrointestinal diseases (Irritable Bowel syndrome, Crohn's disease or Colitis)
* Immune compromised
* Have cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Gut microbiota associated to the synbiotic treatment | 3 months
  Stools samples will be collected and analyzed before and after the intervention and compared between groups

SECONDARY OUTCOMES:
Changes in weight associated to the synbiotic treatment | 3 months
  Weight (kg) will be monitored every 6 weeks
Changes in glucose levels associated to the synbiotic treatment | 3 months
  A1C (Glycated hemoglobin) levels will be monitored every 6 weeks
Changes in body density associated to the synbiotic treatment | 3 months
  body density . A DXA body scan will be performed at the beginning and end of the intervention
Changes in waist circumference associated to the synbiotic treatment | 3 months
  Waist circumference (cm) will be measured every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: eduardo Huarte, PhD, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
Result of the study will be made available to the scientific community trough manuscript publication. Each participant will be assigned a code to maintain patient confidentiality.